CLINICAL TRIAL: NCT00412672
Title: Protective Effect of Coronary Collaterals on Infarct Size in Patients With Acute Myocardial Infarction
Status: Withdrawn | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Christian Seiler, MD, Professor and Co-Chairman of Cardiology, Department of Cardiology, University Hospital, CH-3010 Bern, Switzerland
Other Study IDs: 37/01
Record Dates: First submitted 2006-12-15; First posted 2006-12-18 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Myocardial Infarction
Keywords: Myocardial infarction; contrast echocardiography; collateral circulation
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The hypothesis of the current proposal is that collateral flow is an important determinant of myocardial protection during an ischemic event. Increased collateral flow for any given area at risk will decrease the myocardial damage caused by the occlusion of the infarct related epicardial artery.

It is further hypothesized that myocardial salvage provided by collateral flow will decrease infarct size and this in turn will decrease LV dilatation post-myocardial infarction.

DETAILED DESCRIPTION:
The hypothesis of the current proposal is that collateral flow is an important determinant of myocardial protection during an ischemic event. Increased collateral flow for any given area at risk will decrease the myocardial damage caused by the occlusion of the infarct related epicardial artery.

It is further hypothesized that myocardial salvage provided by collateral flow will decrease infarct size and this in turn will decrease LV dilatation post-myocardial infarction.

The two primary endpoints are infarct size as assessed by increase of biochemical cardiac markers and coronary collateral perfusion index (CPI) as obtained by transthoracic MCE.

Extent of LV remodelling, i.e., LV dilatation as assessed by serial assessment of LV dimension by LV angiogram and/or echocardiography, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute myocardial infarction with electrocardiographic criterion and/or typical history of angina pectoris and planned revascularisation according to the acute myocardial infarction disease management guidelines of the University Hospital Bern. Including both, patients undergoing primary PCI and patients referred for rescue PCI after failed thrombolytic therapy
* Patients > 18 years old of either sex
* Patients who have given informed consent to the study

Exclusion Criteria:

* Patients unable to give informed consent e.g. because of mechanical ventilation
* Patients with cardiogenic shock
* Patients with myocardial infarction secondary to occlusion of a recently revascularized vessel (subacute stent thrombosis)
* Patients with severe arrhythmias
* Patients whose door-to-balloon time exceeds 120 minutes
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute myocardial infarction undergoing primary PCI as reperfusion therapy of a totally occluded coronary artery.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-07

CONTACTS AND LOCATIONS:
Overall Officials: Christian Seiler, Prof., Principal Investigator — University Hospital Bern, Switzerland